CLINICAL TRIAL: NCT05938192
Title: Predictors of Recurrence After Treatment (Surgery Plus Vaccination) of HPV-related Disease of the Female Genital Tract
Brief Title: Multimodality Treatments of HPV-related Lesions of the Female Genital Tract
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: 572020
Record Dates: First submitted 2023-07-03; First posted 2023-07-10 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-09

CONDITIONS: HPV; Cervical Cancer; Cervix Lesion; Vagina Disease
Keywords: hpv
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vaginal Diseases; Papillomavirus Infections | interventions — Vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with HPV-related disease: Patients with HPV-related disease including cervical and vaginal lesions
  Interventions: Procedure: vaccination

INTERVENTIONS:
Procedure: vaccination — Patients will have surgery (followed by vaccination) for managing HPV-related lesions

SUMMARY:
Cervical cancer is one of the most preventable types of cancer, as it develops over an extended period, and its causative agent is well-known. Persistent infection with human papillomavirus (HPV) is the primary factor causing cervical cancer. Generally, persistent HPV infection leads to cervical dysplasia (also known as cervical intraepithelial neoplasia), which can potentially progress to cancer. Although the majority of women with HPV infection will never develop lesions, a relatively high number of women remain at risk of developing cervical dysplasia. Women with cervical dysplasia who receive appropriate follow-up and treatment are at low risk of developing cervical cancer. However, recurrent cervical dysplasia is a well-known risk factor for cervical cancer. Furthermore, recurrent cervical dysplasia can contribute to morbidity, as additional surgical treatments are associated with fertility and obstetric complications in women who wish to preserve their childbearing potential. Against this background, identifying the best treatment modality for patients with cervical dysplasia is of paramount importance.

The management of residual or recurrent dysplasia after primary treatment is often challenging. Moreover, it is important to classify patients based on their risk of having persistent or recurrent dysplasia following initial treatment. Assessing these risk categories is useful in tailoring appropriate surveillance and determining the need for adjunctive treatments. Our research group has estimated the risk of developing persistent or recurrent dysplasia in several investigations, identifying positive surgical margins, surgical techniques, high-risk HPV infection at the time of diagnosis, and HPV persistence as key prognostic factors. Our findings align with a substantial body of literature investigating this issue. However, accurately estimating the risk of persistent or recurrent dysplasia for each individual patient remains challenging.

Similarly, few studies have evaluated the outcomes of patients affected by vaginal intraepithelial neoplasia, and results have been inconsistent. In fact, there is no consensus on the optimal treatment modality for these patients. Treatments have included topical applications of imiquimod or 5-fluorouracil (5-FU), as well as ablative and excisional procedures performed via conventional surgery, electrosurgery, and carbon dioxide laser. The risk of developing invasive vaginal cancer in these patients remains uncertain, with estimates ranging between 2% and 12% in different series. Recently, a multi-institutional Italian study reported that more than 10% of women initially diagnosed with high-grade vaginal intraepithelial neoplasia were found to have occult invasive vaginal cancer at the time of excisional procedures, highlighting the need for histological diagnosis before proceeding with ablative or medical treatments. Additionally, the widespread implementation of HPV vaccination is expected to reduce the risk of recurrence after treatment.

In this context, the investigators aim to evaluate the significance of post-treatment HPV vaccination and other prognostic factors in influencing the risk of persistent or recurrent lesions of the uterine cervix and vagina.

DETAILED DESCRIPTION:
To assess the risk of recurrence in patients with HPV related lesions treated with surgery with or without HPV vaccination

ELIGIBILITY:
Inclusion Criteria:

* Patients with HPV related disease

Exclusion Criteria:

* consent withdrawal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with newly histological diagnosed moderate /severe dysplasia of the uterine cervix and vagina .
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival | 36 months
  time between surgery and first recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Bogani, Principal Investigator — Giorgio Bogani
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No